CLINICAL TRIAL: NCT01880671
Title: Undersökning av ny Behandlingsmetod Vid migränanfall
Brief Title: Evaluation of a New Treatment for Migraine Attacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jan-Erik Juto, Affiliated professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Migraine2013/657-32
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Migraine Medical Device (Experimental)
  Interventions: Device: Migraine Medical Device
- Inactive Migraine Medical Device (Placebo Comparator)
  Interventions: Device: Inactive Migraine Medical Device

INTERVENTIONS:
Device: Inactive Migraine Medical Device
  Arms: Inactive Migraine Medical Device
Device: Migraine Medical Device
  Arms: Migraine Medical Device

SUMMARY:
The purpose of this study is to evaluate the efficacy of a novel therapy for treatment of migraine, pain reduction and relief of associated symptoms during ongoing migraine attacks, and presence of a preventive effect post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects, in otherwise good health, 20 to 55 years of age
* Subjects who meet the ICHD-2 (2nd Edition of The International Headache Classification) criteria for migraine headache
* Subjects with a minimum of 1 migraine attack per month
* Attack duration of 4 to 72 hours
* Normal attack intensity of at least 4 on a 0-10 VAS-scale

Exclusion Criteria:

* Completed heart surgery
* Cardiovascular disease
* Vascular damage on neck vessels
* Disease other than migraine of the CSN
* Severe disease of vital body organs
* Severe psychiatric disorders
* More than 6 migraine attacks per month

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain intensity according to VAS-scales (0-10) | Estimated 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm, Sweden

REFERENCES:
- [Derived] Juto JE, Hallin RG. Kinetic oscillation stimulation as treatment of acute migraine: a randomized, controlled pilot study. Headache. 2015 Jan;55(1):117-27. doi: 10.1111/head.12485. Epub 2014 Dec 29. PMID 25546476